CLINICAL TRIAL: NCT06319079
Title: Effect of Consumption of a Milk Product Designed for Lactating Women on Human Milk Composition and Nutritional Status of Iron and DHA in Infant Red Blood Cells.. Study in a Vulnerable Population.
Brief Title: Effect of Consumption of a Milk Product Designed for Lactating Women on Human Milk Composition
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Desarrollo e Investigaciones Pediátricas Prof. Dr. Fernando E. Viteri (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UCTH 2024
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Lactating Mothers; Infants
Keywords: human milk; vulnerable population; micronutrients; esencial fatty acids; nutritional supplements
MeSH Terms: interventions — Refit milk powder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The powder milk containers (both SMM and commercial milk) will be packaged by Addvance SA (in the Province of Santa Fe), each of the products will have a label that differentiates them but only the company Addvance SA will know that information. In this project, neither the participating mothers, researchers, and technical staff assigned to the project nor the professional who performs the data analysis knows what product each participant will receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Super 1.000 Mamá (Experimental): Breastfeeding mothers who breastfeed their children during the first four months postpartum will receive a fortified powder milk product formulated and designed specifically for this population.
  Interventions: Dietary Supplement: Fortified powder milk
- Leche comercial (Sham Comparator): Breastfeeding mothers who breastfeed their children during the first four months postpartum will receive commercial powder milk.
  Interventions: Other: Powder milk

INTERVENTIONS:
Dietary Supplement: Fortified powder milk — Super 1.000 Mamá It's made up of milk with added vegetable oils, fish oil, carbohydrates from corn, prebiotic fiber (inulin), vitamins, and minerals, with specifically defined proportions. It has medium energy content, is balanced in protein, fats, and carbohydrates, and provides a significant content of both polyunsaturated fatty acids, such as omega-6, and omega-3, and the added docosahexaenoic acid, as recommended by international organizations. The reconstituted 200 ml serving delivers between 20 and 40% of the Daily Reference Intake in critical nutrients for this particular group of people, which include minerals such as calcium, iron, zinc, iodine, and vitamins such as A, D, C, B12 and folic acid. The rest of the vitamins, and minerals are also at the same level, allowing those who consume it to incorporate a large amount of nutrients regularly. Addvance SA, an SME dairy company from the Province of Santa Fe, will carry out the production of this milk.
  Other Names: Super 1.000 Mamá
  Arms: Super 1.000 Mamá
Other: Powder milk — Commercial powder milk constitutes dehydrated commercially available cow's milk, which is fortified with Vitamins A and D by law.
  Other Names: Commercial powder milk
  Arms: Leche comercial

SUMMARY:
Vulnerable populations, who have deficient diets, may produce human milk (HML) that is not adequate in all nutrients and this will have consequences on the growth and development of the child. In 2021 at IDIP, a specific milk product for pregnant and lactating women Super Mil Mamá ( SMM, whole milk powder fortified with multiple vitamins, minerals and DHA ) has been designed and developed as part of a key strategy to incorporate in public policies for the first 1000 days of life. However, the potential benefits of this product have not yet been evaluated at the population level.

The main objective is to evaluate the effect of the consumption of a milk product (SMM) designed for lactating women on the composition of human milk and the nutritional status of iron and DHA in infant red blood cells in a vulnerable population through a randomized, triple-blind, controlled clinical trial.

Specific objectives To compare the concentrations of DHA, Vitamins A, E, and D, Iron, Iodine, Zinc and Calcium in human milk before and after dietary supplementation with SMM.

To compare the concentrations of DHA, Vitamins A, E, D and Zinc in blood and the nutritional status of maternal iron before and after dietary supplementation with SMM.

To analyze the relationship between micronutrients measured in maternal blood and human milk after dietary supplementation with SMM.

To compare the concentrations of micronutrients measured in blood and human milk in women who received SMM and those who received commercial milk (CM) at the end of supplementation.

To compare the iron nutritional status and DHA content in red blood cells of infants of mothers who consumed SMM or LC.

To evaluate the relationship between the concentration of micronutrients in human milk and infant growth during the first six months of life.

ELIGIBILITY:
Inclusion Criteria:

* Women who attend their child's first check-up within the first month of life, who breastfeed their children, and who consume milk regularly.

Exclusion Criteria:

* Women who have had multiple pregnancies, who receive vitamin or mineral supplements that interfere with the results of the study, and/or women with malabsorption diseases.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
breast milk DHA concentration | breast milk DHA concentration will assessed before starting the intervention (one month postpartum) and at the end of it (fourth month postpartum)
  concentration of DHA in breast milk expressed as a percentage of DHA with respect to the total fatty acids contained in the analyzed sample
breast milk Vitamin A concentration | breast milk Vitamin A concentration will assessed before starting the intervention (one month postpartum) and at the end of it (fourth month postpartum)
  Retinol concentration in breast milk expressed in μmol/L and μg/g fat contained in the analyzed sample
breast milk Vitamin E concentration | breast milk Vitamin E concentration will assessed before starting the intervention (one month postpartum) and at the end of it (fourth month postpartum)
  α-tocopherol concentration in breast milk expressed in μmol/L and μg/g fat contained in the analyzed sample
breast milk Vitamin D concentration | breast milk Vitamin D concentration will assessed before starting the intervention (one month postpartum) and at the end of it (fourth month postpartum)
  25-hidroxi vitamin D concentration in breast milk expressed in ng/ml
breast milk Zinc concentration | breast milk Zinc concentration will assessed before starting the intervention (one month postpartum) and at the end of it (fourth month postpartum)
  Zinc concentration in breast milk expressed in mg/dl
breast milk Calcium concentration | breast milk Calcium concentration will assessed before starting the intervention (one month postpartum) and at the end of it (fourth month postpartum)
  Calcium concentration in breast milk expressed in mg/dl
breast milk Iron concentration | breast milk Iron concentration will assessed before starting the intervention (one month postpartum) and at the end of it (fourth month postpartum)
  Calcium concentration in breast milk expressed in mg/dl
breast milk Iodine concentration | breast milk Iodine concentration will assessed before starting the intervention (one month postpartum) and at the end of it (fourth month postpartum)
  Iodine concentration in breast milk expressed in mg/dl

SECONDARY OUTCOMES:
mother red blood cell DHA concentration | mother serum DHA concentration will assessed before starting the intervention (one month postpartum) and at the end of it (fourth month postpartum)
  concentration of DHA in mother red blood cell expressed as a percentage of DHA with respect to the total fatty acids contained in the analyzed sample
mother Vit A concentration | mother Vit A concentration will assessed before starting the intervention (one month postpartum) and at the end of it (fourth month postpartum)
  Retinol concentration in mother serum expressed in μmol/L
mother Vit E concentration | mother Vit E concentration will assessed before starting the intervention (one month postpartum) and at the end of it (fourth month postpartum)
  α-tocopherol concentration in mother serum expressed in μmol/L
mother Vit D concentration | mother Vit D concentration will assessed before starting the intervention (one month postpartum) and at the end of it (fourth month postpartum)
  25-hidroxi vitamin D concentration in mother serum expressed in ng/ml
mother Zinc concentration | mother Zinc concentration will assessed before starting the intervention (one month postpartum) and at the end of it (fourth month postpartum)
  Zinc concentration in mother serum expressed in mg/dl
mother hemoglobin concentration | mother hemoglobin concentration will assessed before starting the intervention (one month postpartum) and at the end of it (fourth month postpartum)
  hemoglobin concentration in mother serum expressed in g/dL
mother serum ferritin concentration | mother serum ferritin concentration will assessed before starting the intervention (one month postpartum) and at the end of it (fourth month postpartum)
  ferritin concentration in mother serum expressed in ng/ml
child hemoglobin concentration | child hemoglobin concentration will assessed before starting the intervention (one month postpartum) and at the end of it (fourth month postpartum)
  hemoglobin concentration in child serum expressed in g/dL
child serum ferritin concentration | child serum ferritin concentration will assessed before starting the intervention (one month postpartum) and at the end of it (fourth month postpartum)
  ferritin concentration in child serum expressed in ng/ml
child red blood cell DHA concentration | child red blood cell DHA concentration concentration will assessed before starting the intervention (one month postpartum) and at the end of it (fourth month postpartum)
  concentration of DHA in child red blood cell expressed as a percentage of DHA with respect to the total fatty acids contained in the analyzed sample

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Desarrollo e Investigaciones Pediátricas (IDIP) - HIAEP Sor María Ludovica, La Plata, Buenos Aires, Argentina